CLINICAL TRIAL: NCT00051415
Title: A Double Blind, Randomized, Placebo Controlled Trial of Flaxseed in Patients With Hypercholesterolemia
Brief Title: Safety and Effectiveness of Flaxseed for Reducing High Cholesterol
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001291-01 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Hypercholesterolemia
Keywords: Flaxseed; Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

INTERVENTIONS:
Behavioral: Flaxseed-supplemented diet

SUMMARY:
Flaxseed, a rich source of fiber, may be a significant component of a cholesterol-reducing diet. The purpose of this study is to evaluate the safety and effectiveness of flaxseed in reducing high cholesterol.

DETAILED DESCRIPTION:
Hypercholesterolemia is an established risk factor for atherosclerotic cardiovascular disease (ASCVD). The National Cholesterol Education Program estimates that 65 million Americans with hypercholesterolemia could be treated with diet and exercise alone. Flaxseed is a potential component of cholesterol-reducing diet regimens. Flaxseed contains significant amounts of soluble fiber and is a rich source of both alpha-linolenic acid and phytoestrogenic ligands, which have been implicated in the prevention of ASCVD. However, flaxseed's phytoestrogenic ligands may have undesirable hormonal effects. This study will systematically evaluate the safety and efficacy of ground flaxseed ingestion in both men and women with hypercholesterolemia.

Participants will be randomized to receive flaxseed or a matching wheat bran control. The test dose of flaxseed will be 40 grams administered in baked products (muffins, bread, or bars). The first 6 study weeks are a diet stabilization phase, followed by a 10-week study phase in which participants are expected to eat two servings of the test food daily. Blood and urine are collected for analysis, which will include measurement of low density lipoprotein cholesterol (LDL-C), post-prandial triglycerides, and urinary isoprostane secretion.

ELIGIBILITY:
Inclusion Criteria

* Men over 45 and post-menopausal women
* LDL cholesterol > 130 mg/dl

Exclusion Criteria

* Established heart, kidney, or liver disease
* Diabetes
* Cancer

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Philippe O Szapary, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States